**PRIVACY ISSUES**: This document contains personal medical information protected by the Privacy Act of 1974 (see AFFIX 33-332) and the Health Insurance Portability and Accountability Act (HIPAA) (see DoD 6025.18-R) and shall be released only as directed by this document.

## INFORMED CONSENT DOCUMENT

81st Medical Group 301 Fisher Street, Room BA144 Keesler AFB MS 39534-2519

# IRB APPROVAL Initial: 25 August 2014

Annual: 19 August 2016 - 1 June 2017

#### TITLE OF STUDY

FKE20140029H, "Short-Term Application of Tocilizumab following Myocardial Infarction (STAT-MI)"

### Principal & Associate Investigator's (Study Doctors) Names, Sqd/Office Symbol, Phone #

| PI – Col Matthew Carroll | 81 MDOS/SGOMJ | 228-376-3829 |
|---------------------------------|------------------|--------------|
| Al – Capt Christopher Smith | 81 MDOS/SGOM | 228-376-3301 |
| Al – Capt Chad Haller | 81 MDOS/SGOM | 228-376-3301 |
| Al – Ms. Audrey Greenwell | 81 MDSS/SGSE | 228-376-4352 |
| Al – Ms. Rishawn Carriere-Ducre | 81 MDSS/SGSE | 228-376-4376 |
| | PURPOSE OF STUDY | |

You are being asked to participate in a research study at the 81st Medical Group, entitled "Short-Term Application of Tocilizumab following Myocardial Infarction (STAT-MI)"

It is anticipated that 125 participants will be enrolled over the next two years. This study will require you have three additional lab tests during your hospitalization, then a final lab test 30 days later and a phone interview to answer a short study questionnaire. Your participation in this research will last a total of 30 days.

#### **PROCEDURES**

As a participant, you will be asked to read, sign, and date this consent form after the study has been verbally explained to you by one of the investigators listed on the front of this form, and all your questions have been answered.

You will undergo the following procedures:

Day of injection (Day 0): Receive the study medication (Tocilizumab) or placebo (saline filled syringe) and have the first lab called a C-Reactive Protein (CRP) (1 tube of blood) drawn. This blood test may be drawn at the time of your other blood tests used to watch and treat your heart attack.

24 hours after injection (Day 1): Have the second lab called a C-Reactive Protein (CRP) (1 tube of blood) drawn.

48 hours after injection (Day 2): Have the third lab called a C-Reactive Protein (CRP) (1 tube of blood) drawn.

Protocol #FKE20140029H PT'S INITIALS\_\_\_\_

\*\*The tracking section below is completed by the Clinical Research Laboratory Staff\*\*

ICD#: \_\_\_\_\_ Date Issued: \_\_\_\_\_ Date Entered in BIRDS/Initials: \_\_\_\_\_

Day 30: Have a final lab called a C-Reactive Protein (1 tube of blood) drawn and undergo a phone interview to answer four questions to see how your health is after receiving the medication.

You will be assigned to one of two treatments by randomization, a process where the treatment you receive is similar to flipping a coin. You will have an equal chance of being assigned to any of the arms.

The treatment of your heart attack will NOT be affected by partaking in this study. In this trial you will get all of the usual drugs and procedures currently accepted as standard or care.

The investigator(s) may use information about your health from your medical records for this study.

Should your physician deem it necessary for you to have a procedure (unrelated to the research study) requiring additional informed consent, a separate informed consent document will be completed at the time of the procedure.

#### RISKS/INCONVENIENCES

The drug that will be studied in this trial is tocilizumab (Actemra). It a medication currently approved for treatment of Rheumatoid Arthritis. It blocks a protein called Interleukin-6 (IL-6). This protein is increased in the first day of a heart attack and remains elevated for several weeks. Higher levels of this protein are associated with worse outcomes in heart attacks.

The most common adverse effects of tocilizumab in clinical studies were infections of the sinuses or lungs, headaches, high blood pressure, and changes in liver blood tests. Swelling, redness, or itching at the place of the injection may also occur. Regular use of tocilizumab has been associated with infections such as tuberculosis and infections of the blood. Tocilizumab may worsen or cause new diseases of the nervous system. Other side effects include reduced levels of white blood cells or platelets as well as rare allergic reactions. In some studies a small tear in the colon was noted in patients who had a condition called diverticulitis.

If you can become pregnant the study investigator will ask for a pregnancy test prior to giving this medication.

A more detailed list of side effects is provided below: (request removal of paragraph above—this is not relevant for the ICD)

Tocilizumab injection data in rheumatoid arthritis (RA) included 2 well designed clinical trials with over 1700 patients watched. A summary of the side effects noted are shown below:

#### **Injection Site Reactions**

Between 2.4 and 10.1% of patients had itching, redness, and/or swelling at the site of the injection of tocilizumab. Most reactions were mild to moderate in severity. Most resolved without any therapy.

## **Immunogenicity**

In the 6-month control period in SC-I, 0.8-1.6% developed anti-tocilizumab antibodies; of these, all developed neutralizing antibodies. No correlation of antibody development to adverse events or loss of clinical response was observed.

(request removal of paragraph above—this is not relevant to this trial)

**Blood Changes:** 

PT'S INITIALS

- A low white blood count was noted in 3.7%. There was no relationship between the low count and infection. Low counts typically go away once the drug has been stopped.
- Up to 5% of patients had a brief, mild increase in liver blood tests. This change seems to happen more with routine use of the drug. These changes typically go away once the medication has been stopped. There is likely little importance to the change as it goes away with stopping the drug.
- An increase in cholesterol may occur, but this may be important with routine use of the
  medication. The importance of this change is not known, but it is probably important when you
  take the drug on a regular basis.

#### BENEFITS

Treatment on this study is an attempt to give you at least as good a chance of preventing further harm 30 days after your heart attack as current medications and interventions. However, There is no guarantee or promise that you will benefit from this study. This study may also benefit others by helping to find out whether this treatment is better than others in treating heart attacks.

#### **ALTERNATIVES**

If you choose not to participate in this study all other treatments currently available to treat your heart attack will be available to you. An additional alternative is to offer no further therapy. You have discussed the risks and benefits of alternative treatment options available with your physician.

Your participation in this study will be completely voluntary. Your decision whether or not to participate will not affect your care at the 81st Medical Group. Your alternative is not to participate in this study.

#### **EVENT OF INJURY**

Your entitlement to medical and dental care and/or compensation in the event of injury is governed by federal laws and regulations. If you have questions about your rights as a research subject you may contact the 81st Medical Group Institutional Review Board at (228) 376-4917.

If you believe you have received a research-related injury you may contact the Director of the Clinical Research Laboratory at (228) 376-3850 or the investigator(s) listed on page 1 of this document.

## OCCURRENCE OF UNANTICIPATED ADVERSE EVENT

If an unanticipated event (clinical or medical misadventure) occurs during participation in this study you will be informed.

#### CONFIDENTIALITY OF RECORDS OF STUDY PARTICIPATION

Record of your participation in this study may only be disclosed in accordance with federal law, including the Federal Privacy Act, 5 U.S.C. Section 552a, and its implementing regulations. DD Form 2005, Privacy Act Statement-Health Care Records, contains the Privacy Act Statement for the records. By signing this document you give permission for information gained from your participation in this study to be published in medical literature, discussed for educational purposes, and used generally to further medical science. You will not be personally identified; all information will be presented as grouped data.

Your research is supported by the Department of Defense Research Oversight and Compliance Division (AFMSA/SGE-C) who may access your records to ensure subject protection, along with the 81st Medical Group Institutional Review Board, the U.S. Food and Drug Administration (FDA), other government agencies, and/or the sponsoring agency or their designee.

| | 3 |
|---------------|---|
| PT'S INITIALS | |

Your identifiable health information is protected by the HIPAA (Health Insurance Portability and Accountability Act) Privacy Rule issued by the Department of Health and Human Services. Except as required by law, we will not be able to disclose this information to anyone other than you without your authorization, by a separate document you have signed or will be asked to sign as to any of your identifiable health information expected to be collected in this study.

Complete confidentiality cannot be promised, particularly for military personnel, because information bearing on your health may be required to be reported to appropriate medical or command authorities.

#### **DECISION TO PARTICIPATE**

The decision to take part in this study is completely voluntary on your part. You may choose not to take part in the study. Or you may withdraw your consent at any time and discontinue further participation in this study. Leaving the study will not affect your medical care or entitlement to care. You can still get your medical care from our institution. No matter what decision you make there will be no penalty to you and you will not lose any benefits to which you are entitled.

You have had an opportunity to ask questions about this study, your participation, and the procedures involved. The study doctor will be available to answer any questions concerning procedures throughout this study. If significant new findings develop during the course of this study that may relate to your decision to continue participation, you will be informed. The study doctor or your primary physician may terminate your participation in this study at any time if he/she feels this to be in your best interest.

You may withdraw your consent at any time by sending a letter to Colonel Matthew B. Carroll, 81 MDOS/SGOMJ, 301 Fisher Street, Room GA144, Keesler AFB MS 39534 to inform him of your decision.

You will not be paid for participating in this study.

ALL subjects will be treated in compliance with all applicable service, DoD and Federal regulations, and all applicable FDA and HHS guidelines.

I have read all of the above. My questions have been answered concerning areas I did not understand. I am willing to take part in this study. After I sign this form, I will receive a copy.

| SUBJECT'S PRINTED NAM | E | DATE/TIME |
|-----------------------|--------------|-----------|
| FMP (if applicable) | SPONSOR SSN# | |
| SUBJECT'S SIGNATURE | | |
| INVESTIGATOR'S SIGNAT | URE | DATE |

Protocol #FKE20140029H (ADULT ICD)

| RINTED NAME OF INVESTIGATOR | | |
|---|---|---|
| /ITNESS' SIGNATURE | PRINTED NAME OF WITNESS | —————————————————————————————————————— |
| Must witness ALL signatures) | | |
| Distribution: (1) Subject: (2) 81 MDSS/SG | SE (Protocol Coordinator); and (3) Principal In | vestigator |